CLINICAL TRIAL: NCT02005809
Title: Clinical Impact of Second-look Endoscopy After Endoscopic Submucosal Dissection of Gastric Neoplasm
Acronym: SLEGD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kosin University Gospel Hospital (Other)
Collaborators: Inje University (Other)
Responsible Party: Principal Investigator, Park Moo In, Department of internal medicine, Kosin University Gospel Hospital, Kosin University Gospel Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2nd look EGD
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Gastric Neoplasms
Keywords: Endoscopic submucosal dissection; gastric neoplasm; second look endoscopy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Second look endoscopy (Active Comparator): This group is performed second look endoscopy about 24 hours later from endoscopic submucosal dissection.
  Interventions: Procedure: second look endoscopy
- without second look endoscopy (No Intervention): This group is not performed second look endoscopy after ESD

INTERVENTIONS:
Procedure: second look endoscopy — Second look endoscopy includes observation or prophylactic bleeding control of ESD site.
  Arms: Second look endoscopy

SUMMARY:
Gastroenterologists often follow up second look endoscopy after endoscopic submucosal dissection(ESD) of gastric neoplasms because they want to prevent bleeding of procedure sites. But Goto suggested in his retrospective analysis that a second-look endoscopy after endoscopic submucosal dissection for gastric epithelial neoplasm may be unnecessary. So, the investigators try to identify the hypothesis prospectively in this study.

ELIGIBILITY:
Inclusion Criteria:

* histological confirmed patients(gastric adenoma or adenocarcinoma)
* performed gastric ESD patients about 24 hours before

Exclusion Criteria:

* perforation after ESD
* piecemeal resection of ESD specimen
* hemostatic agent or proton pump inhibitor users before ESD
* heparin or antiplatelet agent users
* Serious concurrent infection or nonmalignant illness that is uncontrolled
* Psychiatric disorder that would preclude compliance
* Allergy history to proton pump inhibitor

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Post-ESD bleeding rate according to second look endoscopy | Up to 60days

SECONDARY OUTCOMES:
bleeding complication rate according to location of lesion in stomach. | Up to 60days
  Fundus, cardia, upper body, mid body, lower body, antrum anterior wall, posterior wall, great curvature, lesser curvature
Bleeding rate according to size of resected specimen | Up to 60days
  longest diameter of specimen: millimeter
Post ESD bleeding rate according to total procedure time of endoscopic submucosal dissection | Up to 60days
Post ESD bleeding rate according to bleeding degree during endoscopic submucosal dissection | Up to 60days
  Mild: bleeding control time: <1/3 of total ESD procedure time. Moderate: bleeding control time: 1/3~1/2 of total ESD procedure time Severe: bleeding control time: >1/2 of total ESD procedure time

CONTACTS AND LOCATIONS:
Locations (1):
- Kosin University Gospel Hospital, Busan, South Korea

REFERENCES:
- [Background] Ohkuwa M, Hosokawa K, Boku N, Ohtu A, Tajiri H, Yoshida S. New endoscopic treatment for intramucosal gastric tumors using an insulated-tip diathermic knife. Endoscopy. 2001 Mar;33(3):221-6. doi: 10.1055/s-2001-12805. PMID 11293753
- [Background] Takeshita K, Tani M, Inoue H, Saeki I, Honda T, Kando F, Saito N, Endo M. A new method of endoscopic mucosal resection of neoplastic lesions in the stomach: its technical features and results. Hepatogastroenterology. 1997 Nov-Dec;44(18):1602-11. PMID 9427030
- [Background] Goto O, Fujishiro M, Kodashima S, Ono S, Niimi K, Hirano K, Yamamichi N, Koike K. A second-look endoscopy after endoscopic submucosal dissection for gastric epithelial neoplasm may be unnecessary: a retrospective analysis of postendoscopic submucosal dissection bleeding. Gastrointest Endosc. 2010 Feb;71(2):241-8. doi: 10.1016/j.gie.2009.08.030. Epub 2009 Nov 17. PMID 19922919
- [Background] Tsuji Y, Ohata K, Ito T, Chiba H, Ohya T, Gunji T, Matsuhashi N. Risk factors for bleeding after endoscopic submucosal dissection for gastric lesions. World J Gastroenterol. 2010 Jun 21;16(23):2913-7. doi: 10.3748/wjg.v16.i23.2913. PMID 20556838
- [Background] Takizawa K, Oda I, Gotoda T, Yokoi C, Matsuda T, Saito Y, Saito D, Ono H. Routine coagulation of visible vessels may prevent delayed bleeding after endoscopic submucosal dissection--an analysis of risk factors. Endoscopy. 2008 Mar;40(3):179-83. doi: 10.1055/s-2007-995530. PMID 18322872
- [Background] Kim JW, Kim HS, Park DH, Park YS, Jee MG, Baik SK, Kwon SO, Lee DK. Risk factors for delayed postendoscopic mucosal resection hemorrhage in patients with gastric tumor. Eur J Gastroenterol Hepatol. 2007 May;19(5):409-15. doi: 10.1097/MEG.0b013e32801015be. PMID 17413293
- [Background] Uedo N, Takeuchi Y, Yamada T, Ishihara R, Ogiyama H, Yamamoto S, Kato M, Tatsumi K, Masuda E, Tamai C, Yamamoto S, Higashino K, Iishi H, Tatsuta M. Effect of a proton pump inhibitor or an H2-receptor antagonist on prevention of bleeding from ulcer after endoscopic submucosal dissection of early gastric cancer: a prospective randomized controlled trial. Am J Gastroenterol. 2007 Aug;102(8):1610-6. doi: 10.1111/j.1572-0241.2007.01197.x. Epub 2007 Mar 31. PMID 17403076
- [Background] Chung IK, Lee JH, Lee SH, Kim SJ, Cho JY, Cho WY, Hwangbo Y, Keum BR, Park JJ, Chun HJ, Kim HJ, Kim JJ, Ji SR, Seol SY. Therapeutic outcomes in 1000 cases of endoscopic submucosal dissection for early gastric neoplasms: Korean ESD Study Group multicenter study. Gastrointest Endosc. 2009 Jun;69(7):1228-35. doi: 10.1016/j.gie.2008.09.027. Epub 2009 Feb 27. PMID 19249769
- [Background] Gotoda T, Yanagisawa A, Sasako M, Ono H, Nakanishi Y, Shimoda T, Kato Y. Incidence of lymph node metastasis from early gastric cancer: estimation with a large number of cases at two large centers. Gastric Cancer. 2000 Dec;3(4):219-225. doi: 10.1007/pl00011720. PMID 11984739
- [Background] Ono H, Kondo H, Gotoda T, Shirao K, Yamaguchi H, Saito D, Hosokawa K, Shimoda T, Yoshida S. Endoscopic mucosal resection for treatment of early gastric cancer. Gut. 2001 Feb;48(2):225-9. doi: 10.1136/gut.48.2.225. PMID 11156645
- [Background] Fujishiro M, Kodashima S, Goto O, Ono S, Muraki Y, Kakushima N, Omata M. Technical feasibility of endoscopic submucosal dissection of gastrointestinal epithelial neoplasms with a splash-needle. Surg Laparosc Endosc Percutan Tech. 2008 Dec;18(6):592-7. doi: 10.1097/SLE.0b013e318187973f. PMID 19098667
- [Background] Shimatani T, Inoue M, Kuroiwa T, Xu J, Tazuma S, Horikawa Y, Nakamura M. Acid-suppressive efficacy of a reduced dosage of rabeprazole: comparison of 10 mg twice daily rabeprazole with 20 mg twice daily rabeprazole, 30 mg twice daily lansoprazole, and 20 mg twice daily omeprazole by 24-hr intragastric pH-metry. Dig Dis Sci. 2005 Jul;50(7):1202-6. doi: 10.1007/s10620-005-2760-0. PMID 16047460